CLINICAL TRIAL: NCT04497415
Title: The COVID-19 and Healthcare Workers: An Active Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Professor of medical psychology, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 8032
Record Dates: First submitted 2020-08-02; First posted 2020-08-04 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Brief Video-based Intervention; Non Intervention Control

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based intervention (Experimental): A brief video about coping with COVID-19 stress presented to the participants
  Interventions: Other: Video-Based intervention
- Assessment only (No Intervention): Control

INTERVENTIONS:
Other: Video-Based intervention — Three minutes video of a nurse that shares her personal story
  Arms: Video-based intervention

SUMMARY:
The overarching goal of this study is to examine the efficacy of a brief video intervention in reducing stigma and fear, and improving help-seeking behavior, among health care providers (N=1,200), with pre- post- and follow-up assessments (at day 14 and day 30). Participants will be recruited via Amazon Turk and randomly assigned to either a) a video-based intervention (day 1 and a "booster intervention" of the same content on day 14 of the study) featuring the personal story of a health care provider during COVID-19 pandemic, his/her struggles and barriers to care, (b) video-based intervention (day 1 only), and a written description of the same story on day 14 (c) no-intervention control arm (questionnaires only).

The invetsigators aim to (1) determine whether video-based intervention reduce stigma and fear, and increase help-seeking behavior in relation to COVID-19 among health care providers, and (2) compare high-risk areas (e.g., NY) to low-risk areas (e.g., Montana) on intervention outcomes, and (3) test whether symptoms of depression, anxiety, PTSD and Moral Injury (measured by the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder (GAD-7), the Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) and the Moral Injury Events Scale (MIES)) would change over time.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) has widely and rapidly spread around the world. To effectively respond to the COVID-19 outbreak, various governments have implemented rapid and comprehensive public health emergency interventions that include social restrictions and quarantines, which is the separation and restriction of movement of people who might have been exposed to the virus. While the physical risk (e.g. pneumonia, respiratory breakdown) is getting the most scientific and clinical attention, this outbreak also has significant mental health risks and extreme psychological fear-related responses. Psychological responses to previous large-scale outbreaks, particularly to the Ebola Virus Disease (EVD) epidemic during 2014-2016, provide insight into the potential impact of rapidly spreading diseases on mental health problems. During the Ebola outbreak, fear-related behaviors such as stigmatizing infected survivors and ignoring medical procedures impeded public health efforts and negatively affected the recovery of survivors. Anxiety, posttraumatic stress disorder (PTSD), and depression were found in nearly half of the EVD survivors and their contacts.

The COVID-19 outbreak exceeds the scope and magnitude of most previous disasters over the last 100 years. It entails a blend of risk factors for both acute and long-term mental health problems. Data that is started to emerge from the COVID-19 outbreak, suggest that front lines health workers (doctors; nurses) are particularly at risk. A recent study in 1257 health care workers from 34 hospitals, conducted between January 29 to February 3, 2020, revealed that more than half (50.4%) of the health workers were screened positive for depression, 44.6% for anxiety, and 34.0% for insomnia. Consistent with previous disaster studies a dose-response relationship was found between the level of exposure and outcomes. Others may develop a moral injury, profound psychological distress which results in actions, or the lack of them, which violet one's moral or ethical code. Given the magnitude of the COVID-19 outbreak, its risk to physical and mental health, an effective and timely response is essential to address the psychosocial needs associated with the ongoing exposure to disease, death, and distress among health care providers, across low and high risks areas.

Many health care providers reluctant to seek support from friends and family, as well as mental health care due to stigma and fear (e.g., "it would be too embarrassing", "I would be seen as week"). Despite enduring symptoms, they may wait months to years before they seek help. Among reasons to avoid seeking mental health care, individuals report mistrust in mental health providers, being seen as weak or stereotyped as "crazy", and a belief that they may be responsible for having mental health problems. Applying strategies to reduce stigma and fear towards mental health care and improve help-seeking behavior may ameliorate impaired functioning and reduce risks for long-term psychiatric illness.

Previous studies have shown that social contact is the most effective type of intervention to reduce stigma- related attitudes and to improve help-seeking behavior. Social contact involves interpersonal contact with members of the stigmatized group: members of the general public who meet and interact with individuals who suffer from stress, fear, depression, or anxiety and seek mental health care, are likely to lessen their stigma. Corrigan has identified the most important ingredients of contact-based programs: an empowered presenter with lived experience who attains his/her goals (e.g., "I was able to fight the depression/distress that I had following the COVID-19"). While both direct, in-person social contact and indirect, video-based social contact have effectively improved attitudes toward mental issues and care, the latter can be implemented on a larger scale, use a minimal resource and easily disseminated.

ELIGIBILITY:
Inclusion Criteria:

English speakers Healthcare workers aged 18-80 and residents of the USA.

Exclusion Criteria:

Non-English speakers, non-healthcare workers, age less than 18 or more than 80, non-US residents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — Columbia University and NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video-based Intervention | Assessment Only
Started (Pre-intervention assessment (day 1)) | 229 | 121
Post-intervention Assessment (Day 1) | 229 | 121
First Follow-up Assessment (Day 14) | 195 | 102
Completed (Second follow-up assessment (day 30)) | 186 | 94
Not Completed | 43 | 27
Not completed — Lost to Follow-up | 43 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video-based Intervention | Assessment Only | Total
Number analyzed (Participants) | 229 | 121 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (11.5) | 33.8 (11.5) | 34.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 95 | 260
  Male | 64 | 26 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 6 | 34
  Not Hispanic or Latino | 201 | 115 | 316
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 23 | 15 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 15 | 46
  White | 170 | 86 | 256
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 229 | 121 | 350
Occupation [Count of Participants; unit: Participants]
  Nurse | 156 | 81 | 237
  Physician | 37 | 15 | 52
  EMT | 20 | 10 | 30
  Other | 16 | 15 | 31
Exposure to COVID-19 [Count of Participants; unit: Participants] | 105 | 46 | 151

OUTCOME MEASURES:

1. Primary Outcome: Help-seeking Behavior
Description: Measured with the Attitudes Towards Seeking Professional Psychological Help Scale (ATSPPH) - total scores range from 3 to 12, with higher scores indicating greater treatment-seeking intentions
Time Frame: Assessed at baseline and post-intervention (both day 1), first follow-up (day 14), and second follow-up (day 30)
Population: Fifty-three participants were lost to follow-up before first follow-up (day 14) and 70 were lost to follow-up before second follow-up (day 30).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Video-based Intervention | Assessment Only
Number analyzed (Participants) | 229 | 121
units on a scale
  Baseline | 8.2 [7.9 to 8.5] | 8.5 [8.1 to 8.9]
  Post-intervention | 9.3 [9.0 to 9.6] | 8.7 [8.2 to 9.1]
  First follow-up (day 14): number analyzed (Participants) | 195 | 102
  First follow-up (day 14) | 9.7 [9.4 to 10.0] | 9.3 [8.9 to 9.7]
  Second follow-up (day 30): number analyzed (Participants) | 186 | 94
  Second follow-up (day 30) | 9.4 [9.1 to 9.7] | 9.1 [8.8 to 9.5]

2. Primary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: Measured with the GAD-7 scale - total scores range from 0 to 21, with higher scores indicating greater self-reported anxiety
Time Frame: Assessed at baseline, 14-day follow-up, and 30-day follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video-based Intervention | Assessment Only
Number analyzed (Participants) | 229 | 121
units on a scale
  Baseline (day 1) | 7.6 (5.9) | 6.7 (6.1)
  First follow-up (day 14): number analyzed (Participants) | 195 | 102
  First follow-up (day 14) | 6.9 (6.0) | 5.9 (5.2)
  Second follow-up (day 30): number analyzed (Participants) | 186 | 94
  Second follow-up (day 30) | 6.5 (5.7) | 5.4 (5.3)

3. Primary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: Measured with PHQ-9 - total scores range from 0 to 27; higher scores indicate greater self-reported depression
Time Frame: Assessed at baseline, 14-day follow-up, and 30-day follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video-based Intervention | Assessment Only
Number analyzed (Participants) | 229 | 121
units on a scale
  Baseline (day 1) | 7.9 (6.6) | 6.6 (5.6)
  First follow-up (day 14): number analyzed (Participants) | 195 | 102
  First follow-up (day 14) | 7.4 (6.7) | 6.0 (5.7)
  Second follow-up (day 30): number analyzed (Participants) | 186 | 94
  Second follow-up (day 30) | 7.0 (6.2) | 5.4 (5.7)

4. Primary Outcome: Primary Care Posttraumatic Stress Disorder (PC-PTSD) Screen
Description: Measured with the PC-PTSD for DSM-5 - total scores range from 0 to 5, with higher scores indicating greater self-reported PTSD symptoms
Time Frame: Assessed at baseline, 14-day follow-up, and 30-day follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video-based Intervention | Assessment Only
Number analyzed (Participants) | 229 | 121
units on a scale
  Baseline (day 1) | 1.9 (1.6) | 1.8 (1.7)
  First follow-up (day 14): number analyzed (Participants) | 195 | 102
  First follow-up (day 14) | 1.8 (1.6) | 1.2 (1.5)
  Second follow-up (day 30): number analyzed (Participants) | 186 | 94
  Second follow-up (day 30) | 1.7 (1.7) | 1.4 (1.6)

5. Primary Outcome: Moral Injury Events Scale (MIES)
Description: Measured with the MIES - scores range from 9 to 36, with higher scores indicating greater moral injury
Time Frame: Assessed at baseline, 14-day follow-up, and 30-day follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video-based Intervention | Assessment Only
Number analyzed (Participants) | 229 | 121
units on a scale
  Baseline (day 1) | 18.1 (6.4) | 17.1 (6.6)
  First follow-up (day 14): number analyzed (Participants) | 195 | 102
  First follow-up (day 14) | 18.1 (6.8) | 16.5 (6.3)
  Second follow-up (day 30): number analyzed (Participants) | 186 | 94
  Second follow-up (day 30) | 17.5 (6.7) | 16.5 (6.9)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Our definition of adverse event and serious adverse event does not differ from the clinicaltrials.gov definition.
Arm/Group | Video-based Intervention | Assessment Only
All-Cause Mortality (participants affected / at risk) | 0/229 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/229 | 0/121
Other Adverse Events (participants affected / at risk) | 0/229 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT04497415/Prot_SAP_001.pdf